CLINICAL TRIAL: NCT06136377
Title: Evaluation of the Concordance Between Pre-therapy Dosimetry Performed From 68Ga-PSMA-11 Dynamic PET and Post-treatment Dosimetry of 177Lu-PSMA-617 Vectorized Internal Radiotherapy in Patients With Metastatic Prostate Cancer Resistant to Hormonal Castration.
Acronym: GaLuPro
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-A02235-40
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Patients With Metastatic Castration-resistant Prostate Cancer
Keywords: nuclear medicine; prostate cancer; taxane chemotherapy; 68Ga-PSMA-11
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RIV treatment with 177Lu-PSMA-617. (Experimental)
  Interventions: Radiation: 177Lu-PSMA-617 PET scan

INTERVENTIONS:
Radiation: 177Lu-PSMA-617 PET scan — Patients then begin their first course of treatment an average of 2 months after the 68Ga-PSMA-11 PET scan, with IVR usually divided into a total of 6 courses. During the first course of treatment, patients undergo an initial SPECT scan 5h (±1h) post-injection, and return to the nuclear medicine department for three further SPECT scans, at 24h, 4 days and 8 days post-injection.

SUMMARY:
Patients undergo three diagnostic PET scans: 18F-FDG PET scan / 18F-Choline PET scan and 68Ga-PSMA PET scan. Following the diagnostic PET scans, and if patients' eligibility for 177Lu-PSMA-617 IVR treatment is confirmed, SPECT acquisitions will be performed during the first treatment course at 5h, 24h, 4 days and 8 days for dosimetric control.

The patient will then return to the nuclear medicine department to undergo SPECT/CT (3 FOV) acquisitions using the same methods as those presented above and recommended in the standard management at : D+24h post-injection, D+4d post-injection and D+8d post-injection No further research-specific acts or procedures will be performed at the end of the first treatment course.

Continuity of treatment will be carried out in accordance with standard management and treatment requirements and modalities, as will clinical, biological and radiological follow-up.

DETAILED DESCRIPTION:
Internal vectored radiotherapy (IVRT) for mCPRCs is emerging as a new treatment line of choice. Radiolabeled molecules with a high affinity for PSMA have emerged as promising theranostic radiopharmaceuticals for the management of mCPRCs.

The 177Lu-PSMA-617 had substantial anti-tumor effects, including a beneficial effect on survival in cases of mCRPC. With regard to the choice of diagnostic radiopharmaceutical, which must be homologous to the therapeutic agent, 68Ga-PSMA-11 PET/CT showed significantly higher sensitivity and specificity than traditional radiological imaging for detecting lymph node or bone metastases in prostate cancer. The evaluation of 177Lu-PSMA-617 as a new radiopharmaceutical also requires a dosimetry step, which is essential for studying the "injected activity - therapeutic response - adverse effects/toxicity" relationship.

The aim of this study is to carry out a dynamic 68Ga-PSMA-11 PET acquisition in order to evaluate pre-therapy absorbed doses and to compare these with post-therapy dosimetry carried out during the first course of 177Lu-PSMA-617 treatment using SPECT acquisitions.

This research is part of standard management and will not modify the activities of radiopharmaceuticals administered during diagnostic PET examinations with 18F-FDG, 18F-Choline and 68Ga-PSMA-11 or during treatment with 177Lu-PSMA-617.

Patients undergo three diagnostic PET scans: 18F-FDG PET scan / 18F-Choline PET scan and 68Ga-PSMA PET scan. Following the diagnostic PET scans, and if patients' eligibility for 177Lu-PSMA-617 IVR treatment is confirmed, SPECT acquisitions will be performed during the first treatment course at 5h, 24h, 4 days and 8 days for dosimetric control.

The patient will then return to the nuclear medicine department to undergo SPECT/CT (3 FOV) acquisitions using the same methods as those presented above and recommended in the standard management at : D+24h post-injection, D+4d post-injection and D+8d post-injection No further research-specific acts or procedures will be performed at the end of the first treatment course.

Continuity of treatment will be carried out in accordance with standard management and treatment requirements and modalities, as will clinical, biological and radiological follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 with histologically proven metastatic prostate cancer treated with taxane chemotherapy plus at least one second-generation hormone therapy and resistant to hormonal castration (eligibility criterion for 177Lu-PSMA IVR treatment).
* Patient referred to CGFL for standard disease management with indication for 18F-FDG PET, 18F-Choline PET and 68Ga-PSMA-11 PET to validate patient's eligibility for 177Lu-PSMA-617 IVR treatment.
* ECOG ≤ 2
* Life expectancy ≥ 6 months
* No unacceptable medical or radiological risk for isolation in a nuclear medicine therapy unit.
* Patient informed about the study, able to understand the study constraints and sign the consent form.
* Patient affiliated to the social security system or equivalent

Exclusion Criteria:

* Inability of the patient to maintain a lying position, without moving, for more than 1 hour (1 hour 20 minutes of acquisition for the dynamic PET acquisition specific to the GaLuPro study).
* Allergy to 68Ga-PSMA-11 or 177Lu-PSMA-617
* Contraindications to receiving 177Lu-PSMA IVR treatment and/or performing the imaging tests required by the protocol (patient with pacemaker or defibrillator).
* Urinary tract obstruction or hydronephrosis. Patients with a diagnosis or high risk of urinary retention and/or fitted with a urinary catheter and/or with incontinence making urine collection impossible or PET examinations impossible.
* Patient refusal to participate in study
* Impossibility for the patient to undergo medical monitoring and compliance with treatment and trial procedures for geographical, social or psychological reasons.
* Persons deprived of their liberty or under guardianship (including curatorship)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Study the correlation between pre- and post-treatment estimates of absorbed doses to organs at risk | During 12 months
  Pre-treatment absorbed dose estimates will be determined during 68Ga-PSMA-11 PET acquisitions. Post-treatment absorbed dose estimates will be determined using 177Lu-PSMA-617 SPECT acquisitions.

IPD SHARING:
Plan to Share IPD: No